CLINICAL TRIAL: NCT06247423
Title: Effects of 10kHz High-frequency Alternating Current Transcutaneous Stimulation on Tremor in People with Parkinson's Disease
Brief Title: High-frequency Alternating Current Stimulation for Tremor in Parkinson's Disease.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Collaborators: Ministry of Science and Innovation, Spain (Other Government); Asociación Parkinson Toledo (CAP Toledo) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Parkinson-neuromodest-gifto; MCIN/10.13039/501100011033 (Other: Ministery of science and innovation of Spain)
Record Dates: First submitted 2024-01-22; First posted 2024-02-07 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Parkinson's Disease and Parkinsonism; Nerve Block; Motor Activity
Keywords: High-frequency alternating current stimulation; Parkinson's Disease; Tremor; Motor activity
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders; Motor Activity; Tremor

STUDY DESIGN:
Intervention Model Description: Two interventions will be performed:
  * Intervention A: active stimulation (High-frequency current stimulation 10kHz).
  * Intervention B: sham stimulation (simulated electrical stimulation).
Who Masked: Participant, Outcomes Assessor
Masking Description: Blinding of participants will be performed using the same equipment, electrodes, and placement for the real or sham stimulation treatments. In addition, both the participants and the outcome assessor will not have a view of the equipment screen.
  Blinding of the outcome assessor will be performed using different team members for randomization of the interventions (Researcher 1), intervention (Researcher 2), evaluation (Researcher 3), and statistical analysis (Researcher 4). Randomization will be kept hidden from participants and research team members and only the researcher who will deliver the intervention (Researcher 2) will know the group assignment. Successful blinding of participants and evaluator will be analyzed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 10kHz (Experimental): Alternating current stimulation with a 10kHz frequency with a transcutaneous approach, 20 minutes for each intervention.
  Interventions: Device: Active group 10kHz
- Sham stimulation (Sham Comparator): Sham stimulation via transcutaneous approach will be delivered only for the first 30 seconds, following the same procedures as the 10kHz group.
  Interventions: Device: Sham intervention

INTERVENTIONS:
Device: Active group 10kHz — For electrical stimulation in the active groups, unmodulated alternating currents with a symmetrical rectangular waveform of 10 kHz will be applied for 20 minutes. The current intensity shall be adjusted individually for each participant by increasing the current intensity until the participant reports a "strong but comfortable tingling" sensation just below the motor threshold. One electrode will be placed over the median and radial nerves, while the other over the radial nerve.
  The intensity of the current shall be adjusted every two minutes if the tingling sensation decreases. This protocol had been used in previous studies conducted by our research group.
  Arms: 10kHz
Device: Sham intervention — Sham electrical stimulation will be performed with the same equipment, time, and electrodes as in the active groups without the participants and the evaluator having a view of the device screen. The intensity of the current will be increased for 30 seconds until the sensory threshold ("strong but comfortable tingling sensation") will be reached and after that, the intensity will be reduced to 0 milliamperes (mA) with 30 seconds ramp down. Participants will not receive electrical current during the rest of the placebo intervention. This protocol was used in other studies with similar interventions to blind participants.
  Arms: Sham stimulation

SUMMARY:
The goal of this randomized, double-blind, placebo-controlled, crossover study is to test the effectiveness of 10 kilohertz (kHz) high-frequency transcutaneous stimulation for tremor in people with Parkinson's disease. The main questions it aims to answer are:

* Compare the effectiveness between sham stimulation and real stimulation (10kHz) for different types of tremors [rest tremor, postural tremor, kinetic tremor], fine motor skills, and maximal isometric handgrip strength.
* Register adverse events, the blinding success of participants and evaluator, and subjective perception of tremor improvement.

Participants will perform the following tasks in an "off" state (without levodopa and dopamine agonists medication). All of them were performed on the upper limb with more tremor.

* Rest Tremor: Forearm on the armrest, count backward from 100 to 0 as fast as possible for 1 minute and 30 seconds.
* Postural Tremor: Extend the arm parallel to the floor (90º shoulder flexion with the forearm extended) for 30 seconds.
* Kinetic Tremor: Hold a cup by the handle, raise it close to the mouth for 3 seconds, then return to the initial position.
* Fine Motor Skills: Complete the nine-hole peg test, placing pegs into holes as quickly as possible.
* Handgrip Strength: Squeeze the device as strongly as possible for 3 seconds, then rest for 15 seconds.

DETAILED DESCRIPTION:
High-frequency alternating current (HFAC) stimulation involves applying electrical stimulation with a frequency above 1 kilohertz (kHz) to peripheral nerves, inducing immediate, reversible nerve block without causing damage. Studies have shown that frequencies between 10 and 20 kHz reduce maximal isometric grip strength when applied transcutaneously over peripheral nerves, suggesting a partial block of A-alpha fibers, which may help reduce nerve hyperexcitability and motor activity. Tremor-related pathologies, influenced by abnormal muscle activity, significantly impact the quality of life of patients, particularly those with Parkinson's disease (PD), where tremor represents one of the most annoying and disabling symptoms since early stages of the disease.

For these reasons, tremor-related pathologies could benefit from HFAC stimulation. To our knowledge, no studies have applied HFAC stimulation in patients with PD. The main objective of this study is to compare the effectiveness of sham stimulation and real stimulation (10kHz) for tremor [rest tremor, postural tremor, kinetic tremor] in people with PD. Secondary objectives include analyzing the effectiveness of stimulation for fine motor skills and maximal isometric grip strength in people with PD, as well as documenting adverse events and evaluating blinding success.

A double-blind, randomized, crossover-design study will be conducted at the University of Castilla-La Mancha. Two interventions will be performed in people with Parkinson's Disease during "Off" state, randomizing the order: Intervention A: 10kHz stimulation; Intervention B: sham electrical stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a confirmed diagnosis of Parkinson's Disease (PD) by a neurologist or specialist physician, specifically with tremor as defined by the consensual declaration of the "Movement Disorder Society".
* Must possess adequate cognitive capacity to perform the tests and understand all the procedure.
* Tolerance to the application of electrotherapy.

Exclusion Criteria:

* Treatment for tremor suppression (deep brain stimulation or medication within 5 hours).
* Altered sensitivity in the intervention area
* Recent traumatism or surgeries which interfere with the measures
* Presence of pacemakers or other implanted electrical devices
* Tattoos or other external agents in the treatment area
* Comorbidities or conditions affecting tremor or coordination (cerebellar injury)

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2024-02-02 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Resting tremor | Before stimulation (T0), during stimulation [at 10 minutes] (T1), immediately after the end of the stimulation [at 20 minutes] (T2), and 10 minutes after the end of the stimulation [at 30 minutes] (T3).
  The tremor activity will be recorded using surface electromyography, linear and angular accelerations with the "Trigno® Wireless Biofeedback System (SP-W06-017 Delsys Inc. Massachusetts, USA)" device, placing one recording sensors on the muscle surface of the extensor digitorum communis and another on the abductor pollicis brevis muscles. All the tests will be measured with the more tremor-affected hand.
  Specifically, for resting tremor the patient will be at rest with their forearms supported, the wrist free, and the elbow flexed at 90 degrees for 1 minute and 30 seconds, while counting backward from 100 to 0 as quickly as possible. Only the last 30 seconds will be registered.
Postural tremor | Before stimulation (T0), during stimulation [at 10 minutes] (T1), immediately after the end of the stimulation [at 20 minutes] (T2), and 10 minutes after the end of the stimulation [at 30 minutes] (T3).
  This outcome will be recorded using the "Trigno® Wireless Biofeedback System".
  For postural tremor, patients will maintain a posture with flexed shoulders at 90 degrees, extended and pronated forearms, with the wrist in a neutral flexion-extension position for 30 seconds.
Kinetic tremor | Before stimulation (T0), during stimulation [at 10 minutes] (T1), immediately after the end of the stimulation [at 20 minutes] (T2), and 10 minutes after the end of the stimulation [at 30 minutes] (T3).
  This outcome will be recorded using the "Trigno® Wireless Biofeedback System".
  For kinetic tremor, patients will be asked to grasp a cup by the handle, always placed at the same distance on the table, bring it to their mouth, hold it in that position for 3 seconds, and then return it to its initial position. The test will be performed with the more tremor-affected hand.

SECONDARY OUTCOMES:
Fine motor skills-finger dexterity | Before stimulation (T0), during stimulation [at 10 minutes] (T1), immediately after the end of the stimulation [at 20 minutes] (T2), and 10 minutes after the end of the stimulation [at 30 minutes] (T3).
  The fine motor skills will be measured using the "Nine-hole peg test", which is a quantitative and standardized test to measure upper limb function. It involves placing 9 plastic pegs located in a container onto a structure with 9 vertical slots on a table. The test will be performed with the more tremor-affected hand. It won't be allowed to grasp/remove multiple pegs simultaneously. Moreover, the time will start when the subject touches the first peg and ends when the last peg touches the container, and the total time will be recorded in seconds. Additionally, the variable of start time will be added, which measures the time from when the instruction will be given until the subject will reach the first peg.
Maximal isometric grip strength | Before stimulation (T0), during stimulation [at 10 minutes] (T1), immediately after the end of the stimulation [at 20 minutes] (T2), and 10 minutes after the end of the stimulation [at 30 minutes] (T3).
  The maximum isometric grip strength will be measured using a hand grip dynamometer (Grip Strength "T.K.K. 5401 GRIP-D, Takei Scientific Instruments CO., LTD., Shinagawa-ku, Tokyo"). The patient's position will be the same as during the measurement of resting tremor, with the dynamometer held by the evaluator.
  The force will be sustained for 3 seconds in 3 pain-free trials, with 15-20 seconds of rest between each trial. The final force measurement will be the average of the 3 trials.
Blinding success | 10 minutes after the end of the stimulation [at 30 minutes] (T3).
  The success of participant and evaluator blinding will be assessed after the intervention. For this purpose, they will be asked the following question: "What type of treatment do you believe you or the participant received?" with five response options: 1) "I strongly believe that I/he/she received an experimental treatment"; 2) "I somewhat believe that I/he/she received an experimental treatment"; 3) "I strongly believe that I/he/she received a placebo"; 4) "I somewhat believe that I/he/she received a placebo"; 5) "I don't know, I do not answer."
  The blinding of subjects and researchers will be assessed using the James' and Bang's blinding indexes.
Adverse events | 10 minutes after the end of the stimulation [at 30 minutes] (T3) and 24 hours after the stimulation (T4).
  Adverse effects caused by the current in both interventions will be collected using a questionnaire format. This includes items with "Yes/No" response options to assess tingling, numbness, stiffness, heat, heaviness, tightness/contraction, weakness, pain (burning, stabbing, electric, superficial, deep), or other sensations in the hand and intervention area, including skin alterations under the electrodes. The perceived unpleasantness level during the intervention will be also evaluated using a numeric pain rating scale, where 0 corresponded to "none" and 10 to "the maximum possible".
Subjective degree of improvement | 10 minutes after the end of the stimulation [at 30 minutes] (T3).
  To assess the patient's subjective degree of improvement, the Patient Global Impression of Improvement (PGI-I) scale will be used after each intervention. This scale will be utilized to evaluate improvement following treatment using a Likert format ranging from 1 to 7, with 1 being "very much improved" and 7 being "very much worse".

CONTACTS AND LOCATIONS:
Overall Officials: Julio Gómez-Soriano, PhD, Principal Investigator — Toledo Physiotherapy Research Group (GIFTO). Castilla la Mancha University.
Locations (1):
- Universidad de Castilla La Mancha, Toledo, Toledo, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arruda BS, Reis C, Sermon JJ, Pogosyan A, Brown P, Cagnan H. Identifying and modulating distinct tremor states through peripheral nerve stimulation in Parkinsonian rest tremor. J Neuroeng Rehabil. 2021 Dec 25;18(1):179. doi: 10.1186/s12984-021-00973-6. PMID 34953492
- [Background] Jitkritsadakul O, Thanawattano C, Anan C, Bhidayasiri R. Tremor's glove-an innovative electrical muscle stimulation therapy for intractable tremor in Parkinson's disease: A randomized sham-controlled trial. J Neurol Sci. 2017 Oct 15;381:331-340. doi: 10.1016/j.jns.2017.08.3246. Epub 2017 Aug 24. PMID 28991711
- [Background] Contreras VT, Araque W, Delgado VS. Trypanosoma cruzi: metacyclogenesis in vitro--I. Changes in the properties of metacyclic trypomastigotes maintained in the laboratory by different methods. Mem Inst Oswaldo Cruz. 1994 Apr-Jun;89(2):253-9. doi: 10.1590/s0074-02761994000200026. PMID 7885254
- See also: We used the references explained on this page to place the electromyography sensors. — http://seniam.org/